CLINICAL TRIAL: NCT01399606
Title: An Open-label Naturalistic Pragmatic Study to Assess the Long Term Safety of BF2.649 (Pitolisant) in the Treatment of Excessive Daytime Sleepiness (EDS) in Narcolepsy (12 Months Follow-up, Followed by a Prolonged Follow up)
Brief Title: Long Term Open Label Study in Narcolepsy With BF2.649 (Pitolisant)
Acronym: HARMONYIII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P09-10 / BF2.649; 2010-023804-28 (EudraCT Number)
Record Dates: First submitted 2011-06-21; First posted 2011-07-22 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Narcolepsy; Cataplexy
Keywords: Excessive Daytime Sleepiness (EDS); Narcolepsy
MeSH Terms: conditions — Narcolepsy; Cataplexy; Disorders of Excessive Somnolence | interventions — pitolisant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BF2.649 (Experimental)
  Interventions: Drug: BF2.649

INTERVENTIONS:
Drug: BF2.649 — 5,10,20,or 40 mg per day, in a once daily scheme
  Other Names: Pitolisant

SUMMARY:
This is a multicentric International Phase III,Long term open label study(12 months)assessing the long-term safety and efficacy of BF2.649 (Pitolisant)in the treatment of Excessive Daytime Sleepiness (EDS) in narcoleptic patients with or without cataplexy.

DETAILED DESCRIPTION:
In narcoleptic patients, results obtained in the previous studies showed that BF2.649 reduced significantly the diurnal somnolence compared to placebo confirming its wakening effect against EDS and demonstrating its anti-cataplectic effect when administrated on an individual titration scheme established on basis of individual benefit/tolerance ratio.This long-term safety pragmatic study will provide information about long-term treatment of BF2.649, and also allow patients who satisfy of BF2.649 treatment in previous or on-going studies of Bioprojet continuing to benefit this product.This is an open-label, naturalistic pragmatic, prospective longitudinal uncontrolled, multi-centre international trial assessing the safety and effect of long-term therapy of BF2.649 in treatment of excessive daytime sleepiness in narcolepsy, on 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged 18 years old and over.
* Patients with a diagnosis of narcolepsy according to the International Classification of Sleep Disorders (ICSD-2) criteria.
* Patients should have complained of EDS with an ESS score at least 12 (historical assessment).
* Patients having previously participated in and completed a Bioprojet narcolepsy study assessing BF2.649 efficacy (P05-03, P06-06, P07-03 HARMONY I or P07-07 HARMONY II, P09-15 HARMONY I bis) or narcoleptic patients complaining with EDS which in the opinion of the investigator would not be able to participate in a double blind study against placebo but who could benefit from testing a new therapy such as the BF2.649 in an open label study.

or patient receiving BF2.649(Pitolisant) under condition of"ATU nominative" according to the French law (called named temporary authorization of use approved by the Afssaps) for Excessive Daytime Sleepiness associated with narcolepsy.

Exclusion Criteria:

* Patients who have discontinued study treatment during the previous studies due to adverse events related to BF2.649.
* Patients with an untreated sleep apnoea syndrome or who have any other cause of daytime sleepiness
* Patients working in an occupation requiring variable shift work or routine night shifts.
* Psychiatric and neurological disorders, other than narcolepsy/cataplexy, or other problem that in the investigator's opinion would preclude the patient's participation and completion of this trial or comprise reliable representation of subjective symptoms.
* Current or recent (within one year) history of a substance abuse or dependence disorder including alcohol abuse as defined in DSM-IV.
* Other active clinically significant illness, including unstable cardiovascular, or neoplasic pathology which could interfere with the study conduct or counter-indicate the study treatments or place the patient at risk during the trial or compromise the study participation.
* Known history of long QTc syndrome, syncope or arrhythmia or any significant serious abnormality of the ECG (e.g. recent myocardial infarction), or QTc interval strictly higher than 450 ms (electrocardiogram Bazett's corrected QT interval
* Severe Hepatic Impairment or with Severe Renal Impairment, or with any other significant abnormality in the physical examination or clinical laboratory results.
* Known hypersensitivity to the tested treatment including active substance and excipients.
* Participation in an other study - in the 30 days prior to the entry in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-05; Primary Completion 2013-10 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Event (TEAE) | 12 months
  Number of Treatment Emergent Adverse Event (TEAE)

SECONDARY OUTCOMES:
efficacy on EDS as measured by ESS ( Epworth Sleepiness Scale) | 12 months
  change from baseline of the score of Epworth Sleepiness Scale score (ESS) and calculation of the rate of responders defined as a reduction of 3 points of the ESS score from baseline or the normalization of the ESS score at 10 or below

CONTACTS AND LOCATIONS:
Overall Officials: Kati Gutierrez, PharmD, Study Director — Bioprojet
Locations (1):
- CHU Montpellier, Montpellier, France